CLINICAL TRIAL: NCT05935423
Title: Intracoronary Allogenic Umbilical Cord Mesenchymal Stem Cell Reduce Infarct Size, Reverse Remodelling, and Improve Cardiac Function
Brief Title: Umbilical Cord Mesenchymal Stem Cell Improve Cardiac Function on ST-elevation Myocardial Infarction (STEMI) Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Indonesia University (Other)
Collaborators: PT. Prodia Stem Cell Indonesia (Industry)
Responsible Party: Principal Investigator, dr. Dede Moeswir, Sp.PD, KKV, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-02-0150
Record Dates: First submitted 2023-05-28; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: Umbilical Cord Mesenchymal Stem Cell; ST Elevation Myocardial Infarction; Infarct Size; Left Ventricular Ejection Fraction; IL-10; VEGF; Galectin 3; GATA-4; Beclin 1; Major Cardiac Adverse Events
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UC-MSC (Experimental): Patients assigned in UC-MSC intervention group will get Umbilical Cord Mesenchymal Stem Cell transplantation
  Interventions: Biological: Umbilical Cord Mesenchymal Stem Cell transplantation
- Control (No Intervention): Patient assigned in control group doesn't get Umbilical Cord Mesenchymal Stem Cell transplantation. However, they will be fully treated based on European Society of Cardiology (ESC) guidelines

INTERVENTIONS:
Biological: Umbilical Cord Mesenchymal Stem Cell transplantation — 50 million UC MSC will be transplanted 10-15 days after primary PCI
  Arms: UC-MSC

SUMMARY:
The goal of this clinical trial is to learn about the effectiveness of Umbilical Cord Mesenchymal Stem Cell (UC MSC) therapy in patients with STEMI against infarct myocardial size reduction and prevent the incidence of heart failure in the future

DETAILED DESCRIPTION:
Participants who have already done Primary Percutaneous Coronary Intervention (PCI) will be informed about the procedure and risk of this clinical trial. After written consent, 60 participants will be check for their eligibility criteria and randomized into intervention (get UC MSC transplantation) and control group. All participants will be check for their biochemical blood analysis: Interleukin-10 (IL-10), Vascular Endothelial Growth Factor (VEGF), Galectin-3, GATA Binding Protein-4 (GATA-4), and Beclin 1 (1 day before transplantation, 7 dan 14 days after transplantation); infarct size and left ventricular ejection fraction (LVEF) through Cardiac MRI (7-10 days after Primary PCI and 6 months after transplantation) and echocardiography (every month); and major adverse cardiac events/MACE (every month). The result will be access after 6 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with STEMI treated with primary PCI maximum 12 hours after onset of chest pain

Exclusion Criteria:

* Patients with history of coronary artery bypass grafting surgery
* Patients with history of heart failure before admission
* Patients with cardiogenic shock
* Patients with cancer disease
* Patients with malignant arrythmia
* Patients with chronic kidney disease
* Patients with haemostasis disorder
* Patients with infection
* Patients with stroke

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Myocardial infarct size change | 6 months
  Myocardial infarct size change in percentage measure with Cardiac MRI 7-10 days after primary PCI to 6 months after UC-MSC transplantation. The method used by measuring the area of infarction in a series of slices and multiplying the area times the slice thickness to determine a volume.

SECONDARY OUTCOMES:
Left Ventricular Ejection Fraction (LVEF) with Echocardiography | 6 months
  Left Ventricular Ejection Fraction (LVEF) measure with Echocardiography every month within 6 months after UC-MSC transplantation
Left Ventricular Ejection Fraction (LVEF) with Cardiac MRI | 6 months
  Left Ventricular Ejection Fraction (LVEF) measure with Cardiac MRI every month within 6 months after UC-MSC transplantation
Major Cardiac Adverse Event (MACE) | 6 months
  Total death, recurrent myocardial infarction, revascularization with primary PCI or Coronary Artery Bypass Graft (CABG) surgery, stroke, rehospitalisation due to heart failure, haemorrhage and arrythmia malignant assess every months within 6 months after UC-MSC transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Dede Moeswir, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Terashvili M, Bosnjak ZJ. Stem Cell Therapies in Cardiovascular Disease. J Cardiothorac Vasc Anesth. 2019 Jan;33(1):209-222. doi: 10.1053/j.jvca.2018.04.048. Epub 2018 Apr 26. PMID 30029992
- [Background] Madonna R, Van Laake LW, Davidson SM, Engel FB, Hausenloy DJ, Lecour S, Leor J, Perrino C, Schulz R, Ytrehus K, Landmesser U, Mummery CL, Janssens S, Willerson J, Eschenhagen T, Ferdinandy P, Sluijter JP. Position Paper of the European Society of Cardiology Working Group Cellular Biology of the Heart: cell-based therapies for myocardial repair and regeneration in ischemic heart disease and heart failure. Eur Heart J. 2016 Jun 14;37(23):1789-98. doi: 10.1093/eurheartj/ehw113. Epub 2016 Apr 7. PMID 27055812
- [Background] Shen H, Wang Y, Zhang Z, Yang J, Hu S, Shen Z. Mesenchymal Stem Cells for Cardiac Regenerative Therapy: Optimization of Cell Differentiation Strategy. Stem Cells Int. 2015;2015:524756. doi: 10.1155/2015/524756. Epub 2015 Aug 3. PMID 26339251
- [Background] Llano R, Epstein S, Zhou R, Zhang H, Hamamdzic D, Keane MG, Freyman T, Wilensky RL. Intracoronary delivery of mesenchymal stem cells at high flow rates after myocardial infarction improves distal coronary blood flow and decreases mortality in pigs. Catheter Cardiovasc Interv. 2009 Feb 1;73(2):251-7. doi: 10.1002/ccd.21781. PMID 19085935
- [Background] Charles CJ, Li RR, Yeung T, Mazlan SMI, Lai RC, de Kleijn DPV, Lim SK, Richards AM. Systemic Mesenchymal Stem Cell-Derived Exosomes Reduce Myocardial Infarct Size: Characterization With MRI in a Porcine Model. Front Cardiovasc Med. 2020 Nov 16;7:601990. doi: 10.3389/fcvm.2020.601990. eCollection 2020. PMID 33304934
- [Background] Timmers L, Lim SK, Arslan F, Armstrong JS, Hoefer IE, Doevendans PA, Piek JJ, El Oakley RM, Choo A, Lee CN, Pasterkamp G, de Kleijn DP. Reduction of myocardial infarct size by human mesenchymal stem cell conditioned medium. Stem Cell Res. 2007 Nov;1(2):129-37. doi: 10.1016/j.scr.2008.02.002. Epub 2008 Mar 8. PMID 19383393
- [Background] Gao LR, Chen Y, Zhang NK, Yang XL, Liu HL, Wang ZG, Yan XY, Wang Y, Zhu ZM, Li TC, Wang LH, Chen HY, Chen YD, Huang CL, Qu P, Yao C, Wang B, Chen GH, Wang ZM, Xu ZY, Bai J, Lu D, Shen YH, Guo F, Liu MY, Yang Y, Ding YC, Yang Y, Tian HT, Ding QA, Li LN, Yang XC, Hu X. Intracoronary infusion of Wharton's jelly-derived mesenchymal stem cells in acute myocardial infarction: double-blind, randomized controlled trial. BMC Med. 2015 Jul 10;13:162. doi: 10.1186/s12916-015-0399-z. PMID 26162993
- See also: Timing of intracoronary bone-marrow-derived stem cell transplantation after ST-elevation myocardial infarction. — https://www.nature.com/articles/ncpcardio0417
- See also: A randomized, open-label, multicenter trial for the safety and efficacy of adult mesenchymal stem cells after acute myocardial infarction. — https://jkms.org/pdf/10.3346/jkms.2014.29.1.23